CLINICAL TRIAL: NCT06006663
Title: Antimicrobial Efficacy of Synthetic Versus Herbal Intracanal Medicaments Against Enterococcus Faecalis
Brief Title: Effect of Hebal and Synthetic Medicamentss on Enterococcus Feacalis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Essam Ahmed Abo Laimon, Demonstrator , Endodontic department,Faculty of dentistry,Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eliminations of E.faecalis
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Effective Intracanal Medicaments Against Enterococcus Faecalis
MeSH Terms: interventions — Ibuprofen; Clindamycin; Ciprofloxacin; Metronidazole; Curcumin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Active Comparator): ibuprofen as intracanal medicament
  Interventions: Drug: Ibuprofen 400 mg.
- group 2 (Active Comparator): modified triple antibiotic paste as intracanal medicament
  Interventions: Drug: modified triple antibiotic paste
- group 3 (Active Comparator): curcumin as intracanal medicament
  Interventions: Dietary Supplement: curcumin
- group 4 (Active Comparator): olive leaves as intracanal medicament
  Interventions: Dietary Supplement: olive leaves extract

INTERVENTIONS:
Drug: Ibuprofen 400 mg. — synthetic intracanal medicament
  Arms: group 1
Drug: modified triple antibiotic paste — synthetic intracanal medicament
  Other Names: clindamycin, ciprofloxacin and metronidazole
  Arms: group 2
Dietary Supplement: curcumin — herbal intracanal medicament
  Arms: group 3
Dietary Supplement: olive leaves extract — herbal intracanal medicament
  Arms: group 4

SUMMARY:
this study aims to evaluate the antimicrobial efficacy of two synthetic (Ibuprofen, Modified triple antibiotic paste) and two herbal materials (Curcumin and Olive leaves extract) used as intracanal medication, against E.Faecalis in secondary endodontic infection cases.

DETAILED DESCRIPTION:
we evaluate the antimicrobial efficacy of two synthetic (Ibuprofen, Modified triple antibiotic paste) and two herbal materials (Curcumin and Olive leaves extract) used as intracanal medication, against E.Faecalis in secondary endodontic infection cases by taking three samples from root canal , the first sample after removing gutta percha from root canal system, the second sample after shaping with protaper universal files and cleaning with 2.5% sodium hypochlorite , the third sample after 7 days from application of the medication .

samples will be diluted into ten fold serial dilution and then the diluted samples will be cultured on bile esculin agar as it is selective media for enterococcus feacalis.

bacterial reduction will be determined and comparision will be made .

ELIGIBILITY:
Inclusion Criteria:

* Single rooted teeth.
* Teeth have clinical signs and symptoms of endodontic failure as sensitivity to percussion, pain, swelling or fistula.
* Teeth with radiographic features of endodontic failure as persistent periapical lesion or widening of periodontal ligament.

Exclusion Criteria:

* • Teeth with fractures of the crown or root.

  * Teeth with periodontal pocket deeper than 4mm.
  * Teeth have procedural error like ledge, broken instrument, or perforation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-26 (Estimated); Primary Completion 2023-10-05 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
measurment of microbial reduction as result of applying synthetic and herbaal intracanal medicaments | time necessary for incubation of each sample is 24 hour
  sample 1 will be taken after gutta percha removal sample 2 will be taken after cleaning and shaping sample 3 will be taken after apllying the intracanal medicament for one week